CLINICAL TRIAL: NCT04831424
Title: The Mitochondrial Stress, Brain Imaging, and Epigenetics Study
Brief Title: Mitochondrial Stress, Brain Imaging, and Epigenetics
Acronym: MiSBIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Dartmouth College (Other); Centre National de la Recherche Scientifique, France (Other); Massachusetts General Hospital (Other); Technische Universität Dresden (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martin Picard, Associate Professor of Behavioral Medicine (in Psychiatry and Neurology), Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NYSPI 7424; 5R01MH122706 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Mitochondrial Diseases
Keywords: Mitochondria; Brain Imaging; Psychophysiology; Epigenetics; Stress; Metabolic rate; Mitochondrial function
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: All participants will undergo TSST and have samples With DNA collected (blood plasma and serum, purified leukocytes, saliva, urine, buccal epithelial cells, hair are stored).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy controls (Experimental): No diagnosis of mitochondrial disease
  Interventions: Behavioral: Trier social stress test
- Mutation (Experimental): Participants carrying the m.3243A>G point mutation, without a diagnosis of MELAS (mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes)
  Interventions: Behavioral: Trier social stress test
- Mutation with MELAS (Experimental): Participants carrying the m.3243A>G point mutation, with a diagnosis of MELAS (mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes)
  Interventions: Behavioral: Trier social stress test
- Deletion (Experimental): Participants carrying a single, large-scale mtDNA deletion
  Interventions: Behavioral: Trier social stress test

INTERVENTIONS:
Behavioral: Trier social stress test — The Trier social stress test (TSST) is a tool for investigating psychobiological stress responses in a laboratory setting. It is a laboratory procedure used to reliably induce stress in human research participants. The study is not examining or validating the test itself but rather using it as a tool to measure the response/focus of study.
  Other Names: TSST

SUMMARY:
The MiSBIE study collects biological, behavioral, psychosocial, neuropsychological, and brain imaging data in participants with either: normal mitochondrial function, individuals with the m.3243A>G mitochondrial DNA (mtDNA) mutation, and individuals a single large-scale mtDNA deletion. These defects induce mitochondrial allostatic load (MAL). The 2-day protocol, plus home-based data collection, will provide a comprehensive assessment of the multi-systemic dysregulation associated with MAL or mitochondrial dysfunction, and the link to physical and mental health-related symptoms.

Aim 1: Determine the influence of MAL on systemic AL biomarkers.

Aim 2: Establish the influence of MAL on stress reactivity profiles.

Aim 3. Examine the association between MAL and psychological functioning.

DETAILED DESCRIPTION:
Age-related physical and cognitive decline, as well as the risk of neurological diseases, are increased by the effects of psychosocial stress. Psychosocial stress triggers neuroendocrine, metabolic, cardiovascular, and inflammatory changes in the body. These changes vary in nature and magnitude between individuals, and are associated with long-term disease risk. However, the biological determinants of the stress response are not well understood.

This project aims to translate the preclinical findings (how mitochondria regulate the different organ systems and major stress response axes are activated during psychological stress) by studying a population of individuals with varying degree of mitochondrial dysfunction, and to test potential neural mechanism, and why some individuals respond more strongly than others to the same stressor.

Each participant will be studied over two consecutive days. Participants will be housed on campus to standardize study conditions. On Day 1, participants will donate blood and saliva, undergo a neuropsychological assessment, and complete questionnaires to assess psychosocial functioning and psychiatric symptoms. After lunch, the investigator will monitor dynamic changes in mental health-related biological outcomes (positive and negative affect, circulating levels of the inflammatory cytokine IL-6, and salivary cortisol) in response to a standardized laboratory challenge. On Day 2, participants will undergo a medical evaluation to assess clinical symptoms and undergo a whole brain neuroimaging session where both resting and stress elicited activity will be measured. A variant of the same stressor as on Day 1 will be used in the neuroimaging session. Participants will then be debriefed, concluding the individuals participation in the study. Participants also complete a home-based saliva and stool collection to examine diurnal variation in salivary hormones, and to examine microbiome composition. This translational project will generate a unique combination of complimentary molecular, cellular, and neuroimaging data that will advance our understanding of the links between mitochondria, the brain, and mental health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women patients between 18 and 55 years of age
* Willing to provide saliva samples and have venous catheter installed for blood collection during the hospital visit
* Willing to provide informed consent and capacity to consent
* Use of effective method of birth control for women of childbearing capacity
* English Speaking

Exclusion Criteria:

* Individuals with cognitive deficit incapable of providing informed consent will not be included
* Symptoms of flu or other seasonal infection four weeks preceding hospital visit
* Raynaud's syndrome (Raynaud phenomenon)
* Involvement in any therapeutic trials listed on clinicaltrials.gov, including exercise
* Metal inside or outside the body or claustrophobia prohibitive to MRI testing
* Diagnosed with mitochondrial disease m.3243A>G, or large scale mtDNA deletion (for healthy controls)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Picard, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be deposited to the NIMH Data Archive.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available at the end of the study, without a expiry date.
Access Criteria: Access will be handled through the NIMH Data Archive (NDA)
URL: https://nda.nih.gov

REFERENCES:
- See also: Study Brochure — http://www.picardlab.org/uploads/7/7/8/4/77845210/1_misbie_brochure_2018-06-26.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
Started | 70 | 20 | 15 | 5
Completed | 70 | 20 | 15 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS | Total
Number analyzed (Participants) | 70 | 20 | 15 | 5 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.6) | 34.4 (11.2) | 43.1 (9.8) | 39.2 (7.6) | 37.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 15 | 11 | 2 | 76
  Male | 22 | 5 | 4 | 3 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 1 | 0 | 10
  Not Hispanic or Latino | 62 | 19 | 14 | 5 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 1 | 0 | 0 | 11
  White | 47 | 18 | 12 | 5 | 82
  More than one race | 2 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 6 | 0 | 1 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 70 | 20 | 15 | 5 | 110

OUTCOME MEASURES:

1. Primary Outcome: Average TSST-induced Elevation in Cortisol
Description: This is designed to measure cortisol reactivity to the trier social stress test (TSST), quantified from salivary cortisol (LC-MS) over an 8-timepoints timecourse. The elevation will be measured as the area under the curve (AUC) for the cortisol time course.
Time Frame: Day 1 post challenge (approximately 2 hours)
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
Number analyzed (Participants) | 70 | 20 | 15 | 5
ng*min/mL | 37.44 (114.60) | 33.86 (54.46) | 42.83 (35.83) | 45.42 (43.65)

2. Primary Outcome: Average Allostatic Load Index
Description: Groups will be compared on a quantitative allostatic load (AL) index integrating baseline fasting measures of neuroendocrine, immune and metabolic systems, urinary catecholamines, hematological measures, and hair/diurnal cortisol levels. 32 different biomarkers were analyzed for this outcome. The full range of the allostatic load index score is 0 to 32. A lower score is considered better, and a higher score is considered worse.
Time Frame: Blood collected on Day 1
Measure: Mean (Standard Deviation); unit: allostatic load score
Arm/Group | Healthy Controls | Mutation | Mutation With MELAS | Deletion
Number analyzed (Participants) | 70 | 20 | 15 | 5
allostatic load score | 9.10 (3.81) | 10.74 (4.05) | 11.31 (3.61) | 12.00 (4.08)

3. Secondary Outcome: Average TSST-induced Elevation in Heart Rate
Description: Groups will be compared on heart rate (HR) as a measure of cardiovascular reactivity to stress, monitored using a continuous 3-lead ECG. The elevation will be computed from the baseline HR to the peak HR reached during the TSST.
Time Frame: Baseline and 2 hours post challenge on Day 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
Number analyzed (Participants) | 70 | 20 | 15 | 5
beats per minute | 14.8 (12.4) | 12.4 (10.7) | 10.9 (6.41) | 12.7 (10.1)

4. Secondary Outcome: Correlation Between Anxiety and Mitochondrial Respiration
Description: The association between mitochondrial respiration using extracellular flux analysis (Seahorse) on blood lymphocytes, and anxiety symptoms measured using the state and trait anxiety inventory (STAI), will be quantified by a linear regression across all study participants.
Time Frame: Day 1
Measure: Number; unit: coefficient of determination (R^2)
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
Number analyzed (Participants) | 70 | 20 | 15 | 5
coefficient of determination (R^2)
  Correlation between mitochondrial respiration and state anxiety | 0.10 | 0.04 | 0.01 | 0.22
  Correlation between mitochondrial respiration and trait anxiety | 0.04 | 0.003 | 0.334 | 0.02

5. Secondary Outcome: Average Neuropsychological Function
Description: The fluency/initiation domain of executive functioning was assessed using the Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test, specifically Condition 1: Letter Fluency total correct. Raw scores were converted to Z-scores based on the control group. A Z-score of 0 represents the mean of the control group, with positive values indicating better performance and negative values indicating worse performance.
Time Frame: Day 2 neuropsychological session
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
Number analyzed (Participants) | 70 | 20 | 15 | 5
Z-score | 0.00 (1.0) | -0.14 (0.96) | -0.58 (1.35) | -0.26 (1.52)

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Healthy Controls | Mutation | Deletion | Mutation With MELAS
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/20 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/20 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/70 | 0/20 | 0/15 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT04831424/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT04831424/SAP_001.pdf